CLINICAL TRIAL: NCT06894485
Title: Effectiveness of Sensory Training in Distal Radius Fractures: A Randomized Controlled Trial
Brief Title: Sensory Training in Distal Radius Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Tugba Civi Karaaslan, Asst. Prof. Dr., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulUr
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Distal Radius Fractures
Keywords: Distal Radius Fractures; Sensory; Physiotherapy; Rehabilitation
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): * Conventional range of motion (ROM) exercises
  * Muscle strengthening exercises
  * Fine motor skill exercises
  * Functional rehabilitation exercises The group will be followed 3 times per week for 8 weeks.
  Interventions: Other: Conventional therapy
- Experimental (Experimental): * Conventional range of motion (ROM) exercises
  * Muscle strengthening exercises
  * Fine motor skill exercises
  * Functional rehabilitation exercises
    • Experimental Group: (Conventional therapy + Sensory Training)
  * Desensitization training (exposure to various textures and stimuli to improve sensory tolerance)
  * Proprioceptive exercises (closed-eye position sense training, weight transfer exercises)
  * Tactile stimulation The group will be followed 3 times per week for 8 weeks.
  Interventions: Other: Conventional therapy; Other: Sensory Training

INTERVENTIONS:
Other: Conventional therapy — * Conventional range of motion (ROM) exercises
  * Muscle strengthening exercises
  * Fine motor skill exercises
  * Functional rehabilitation exercises
Other: Sensory Training — * Desensitization training (exposure to various textures and stimuli to improve sensory tolerance)
  * Proprioceptive exercises (closed-eye position sense training, weight transfer exercises)
  * Tactile stimulation
  Arms: Experimental

SUMMARY:
This randomized controlled trial examines the effectiveness of sensory training in patients undergoing rehabilitation for distal radius fractures. Forty-four participants (aged 18-65, with no prior upper extremity injuries) will be randomly assigned to a control group (conventional physiotherapy) or an experimental group (conventional physiotherapy plus sensory training, including desensitization and proprioception exercises). Assessments will be conducted at baseline, 4 weeks, and 8 weeks using grip strength, sensory function, fine motor skills, pain level, and functional capacity measures. The study aims to compare the impact of sensory training versus conventional physiotherapy on pain reduction, sensory recovery, grip strength, and functional hand use.

DETAILED DESCRIPTION:
This study aims to investigate the effectiveness of sensory training in patients with distal radius fractures. Designed as a randomized controlled trial, the study will include 44 participants aged 18-65 years who have not had a prior upper extremity injury and are in the rehabilitation phase after a fracture. Participants will be randomly assigned to either the control group (receiving conventional physiotherapy) or the experimental group (receiving conventional physiotherapy plus sensory training, including desensitization and proprioception exercises).

Assessments will be conducted before treatment, at 4 weeks, and at 8 weeks. The evaluation tools will include grip strength (hand dynamometer & pinch meter), sensory function (monofilament test), fine motor skills (Nine-Hole Peg Test - NHPT), pain level (Numerical Pain Rating Scale - NPRS), and functional capacity (DASH questionnaire).

The aim of this study is to compare the effects of sensory training versus conventional physiotherapy on pain reduction, sensory recovery, grip strength, and functional hand use.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Diagnosed with distal radius fracture
* In the rehabilitation phase after fracture healing
* No prior upper extremity injuries
* No neurological or psychiatric disorders affecting hand function
* Able to comply with the rehabilitation program

Exclusion Criteria:

* Any other musculoskeletal injury affecting the upper limb
* Previous upper extremity surgeries
* Severe neuropathy or sensory disorders
* Uncontrolled chronic pain conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Monofilament Test | on the first day, four and eight week change
  The monofilament test is a clinical assessment method used to evaluate sensory function and detect peripheral nerve damage. It is widely used in physiotherapy and neurology to measure tactile sensitivity and identify sensory impairments.
  1. The patient is comfortably seated, and the test area is exposed.
  2. Applying the monofilament:
     * The monofilament is placed perpendicularly to the skin surface.
     * It is gently pressed until it reaches its bending point (held for approximately 1-2 seconds).
  3. Patient response: The patient is asked to indicate when they feel the touch.
  4. Recording results: The areas where the patient does or does not feel the stimulus are noted, creating a sensory map.
Numerical Pain Rating Scale | on the first day, four and eight week change
  The Numeric Pain Rating Scale (NPRS) is a measurement method based on the patient's numerical expression of pain. It is commonly used to determine the intensity of pain and track changes during the treatment process.
  Test Procedure Explaining the Scale to the Patient: A scale ranging from 0 to 10 is shown to the patient. 0 = No pain, 10 = The most intense pain imaginable. The patient is asked to choose the number that best represents their current pain.

SECONDARY OUTCOMES:
Grip Strength | on the first day, four and eight week change
  Hand Dynamometer: The hand dynamometer is a device used to measure hand grip strength and is commonly used in the evaluation of hand functions.
  * The device is placed on a stable surface and calibrated to ensure accurate measurement.
  * The patient should sit or stand in a comfortable position, with the elbow typically bent at a 90-degree angle.
  * The patient holds the dynamometer and is asked to squeeze the handle.
  Pinch Meter: Pincer Meter is a device used to measure the strength of a pinching or gripping action, typically between the thumb and index finger.
  * The patient should be seated comfortably or standing, with their elbow typically at a 90-degree angle.
  * The device measures the force exerted between the thumb and index finger.
  * The test will repeat three times, and the highest value is recorded.
Nine-Hole Peg Test | on the first day, four and eight week change
  Nine-Hole Peg Test (9-HPT) is a test used to assess hand function, fine motor skills, and hand coordination. It is commonly used in neurological conditions, hand injuries, and rehabilitation processes.
  Procedure:
  1. Preparation: A pegboard with 9 holes is placed on a flat surface, with a peg in each hole. The patient sits comfortably, and the test is performed on one hand at a time.
  2. Test Execution:
     * Starting Position: The patient prepares by looking at the pegs placed in the starting position.
     * Placing the Pegs: The patient is instructed to pick up each peg and place it into the holes one by one.
     * Test Duration: The time taken to place and remove the pegs is recorded. The test is repeated on both hands.
  3. Results Evaluation: At the end of the test, the total time taken is recorded and used to evaluate hand function. The test is typically repeated three times, and the average time is calculated.
Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire | on the first day, four and eight week change
  The DASH Scale (Disabilities of the Arm, Shoulder, and Hand) is a widely used and valid questionnaire for assessing upper extremity function.
  The DASH scale consists of 30 questions. These questions cover the difficulties patients experience with arm, shoulder, and hand functions, the level of pain they experience, and any difficulties they encounter in daily activities. Additionally, a 5-point Likert scale is used to assess the severity of the complaints (1 = no difficulty, 5 = very difficult).
  Each response is scored, and a total result is obtained. The scores are then evaluated on a scale of 0-100. Lower scores indicate less disability, while higher scores indicate greater functional impairment.
  Evaluation: The results are used to assess the patient's overall functional status and their response to treatment. Higher scores indicate significant difficulties with upper extremity function.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Muurling M, Lotters FJB, Geelen JE, Schouten AC, Mugge W. A long-term effect of distal radius fracture on the sensorimotor control of the wrist joint in older adults. J Hand Ther. 2021 Oct-Dec;34(4):567-576. doi: 10.1016/j.jht.2020.07.002. Epub 2020 Jul 29. PMID 32893099